CLINICAL TRIAL: NCT03010098
Title: The Effect on the Older's Cognition of Dual-loop Target Controlled Infusion Guided by Narcotrend Index
Acronym: POCD;TCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, associate chief physician, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: double closed-loop and POCD
Record Dates: First submitted 2016-12-20; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Anesthesia
Keywords: POCD; narcotrend; closed-loop of target controlled infusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dual-Loop TCI (Experimental): the investigator modified the effect-site target concentrations by NI.If NI fall down to 46 and keep 46 more than 30 seconds,propofol and remifentanil were infused as feedback automatically to achieve the target NI of 26-46.Take blood sample before and after surgery to measure the levels of protein S100beta and NSE.
  Interventions: Device: Dual-Loop TCI
- Open-Loop TCI (Experimental): the investigator modified the effect-site target concentrations of both drugs without minimum or maximum concentration limits without using the Narcotrend monitor only depend on the experience of anesthesiologist.Take blood sample before and after surgery to measure the levels of protein S100beta and NSE.
  Interventions: Device: Open-Loop TCI

INTERVENTIONS:
Device: Dual-Loop TCI — the investigator modified the effect-site target concentrations by NI.If NI fall down to 46 and keep 46 more than 30 seconds,propofol and remifentanil were infused as feedback automatically to achieve the target NI of 26-46
  Other Names: Dual-Loop Target Controlled Infusion of Propofol and Remifentanil Guided by Narcotrend Inde
  Arms: Dual-Loop TCI
Device: Open-Loop TCI — the investigator modified the effect-site target concentrations of both drugs without minimum or maximum concentration limits without using the Narcotrend monitor only depend on the experience of anesthesiologist.
  Other Names: Control infusion of propofol and remifentanil guided by experience
  Arms: Open-Loop TCI

SUMMARY:
To investigate the effect on older's cognition of the application of closed target-controlled infusion(TCI) of propofol and remifentanil guided by Narcotrend index .

DETAILED DESCRIPTION:
Two hundreds of patients scheduled for surgery under general anesthesia were randomly divided into two groups:closed-loop (group A,n=100) and open-loop group(group B,n=100).The procedure during induction of anesthesia was same in two groups.In group A,if Narcotrend index(NI) fall down to 46 and keep more than 30 seconds,propofol and remifentanil were intravenously infused as feedback automatically to achieve the target NI of 26-46.However,the NI in group B was controlled manually.Taking an exam of MMSE before and after the surgery which measures if the older's cognition changed. Furthermore.we will measure the levels of protein S100beta and NSE.

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅰ ~ Ⅱ women undergoing Laparoscopic surgery.
2. Written informed consent from the patient or the relatives of the participating patient.
3. BMI:18.0～25 kg/m2

Exclusion Criteria:

1. Mental illness can not match
2. epidural anesthesia contraindicated
3. People who have Slow-type arrhythmias
4. Chronic renal failure
5. Alcohol or drug abuse
6. Already taking gabapentin, pregabalin, benzodiazepin or antidepression dru

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
MMSE scores | up to 1 week
  The Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment.It is commonly used in medicine and allied health to screen for dementia. It is also used to estimate the severity and progression of cognitive impairment and to follow the course of cognitive changes in an individual over time; thus making it an effective way to document an individual's response to treatment. The MMSE's purpose has been not, on its own, to provide a diagnosis for any particular nosological entity.We measure the patient before the operation and the first/third/seventh day after the operation.

SECONDARY OUTCOMES:
protein s100beta | up to 24 hours
  The calcium-binding protein S100b is enriched in astroglial cells and can cross the blood-brain barrier after hypoxic damage of the central nervous system. Its routine measurement is simple and relatively inexpensive. S100b is filtrated by the kidney and has an estimated half-life of 2 h . Its serum level increases after CA, and its prognostic value has been studied . Because of mitigated results, its routine use has been, up to now, not recommended. S100bata is normally 0.2μg/L in serum or more smaller.We decide to take the blood sample before the operation and after the operation when the patient is awake.

OTHER OUTCOMES:
NSE | up to 24 hours
  NSE has a role in glucose metabolism. As for S100b, NSE is released from the hypoxic brain into the bloodstream, and its serum level correlates with the extent of brain injury. Also, NSE correlates with other markers of brain injury . NSE has a high specificity to predict adverse outcomes when measured in the few days post CA. A cutoff point of 33 mg/l is recommended.in our study, we take the blood sample before the operation and after the operation when the patient awake.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided